CLINICAL TRIAL: NCT02123329
Title: Assessing the Effectiveness of a Pharmacist-delivered Smoking Cessation Program in the State of Qatar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qatar University (Other)
Collaborators: Hamad Medical Corporation (Industry)
Responsible Party: Principal Investigator, Dr. Maguy El Hajj, Assistant Professor and Chair/ Clinical Pharmacy and Practice Section, Qatar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NPRP 4 - 716 - 3 - 203
Record Dates: First submitted 2014-04-20; First posted 2014-04-25 (Estimated); Results first posted 2018-01-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-06

CONDITIONS: Smoking Cessation
Keywords: Qatar; Pharmacy; Pharmacist; Smoking cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control arm (Active Comparator): Participants in the control group will receive 5-10 minutes of unstructured brief smoking cessation advice by the pharmacist. In addition they will be provided with educational materials about smoking cessation and will be offered nicotine replacement therapy (NRT).
  Interventions: Other: Control arm (i.e: regular care)
- Intervention arm (Experimental): Participants assigned to the intervention arm will participate in a face-to-face 4-session program at the pharmacy delivered by the study pharmacist at 2-4-week intervals over 8 weeks in addition to nicotine replacement therapy. The sessions will be set at a date and time that is convenient for both the pharmacist and the participant. The pharmacist will deliver the program at a time different from his or her pharmacy duty regular time.
  Interventions: Behavioral: Pharmacist delivered smoking cessation program

INTERVENTIONS:
Behavioral: Pharmacist delivered smoking cessation program — The first session will be time-intensive taking around 30 minutes. In this session, the study pharmacist will facilitate the participant's preparation to quit. The participant will select a quit date within the next 2-4 weeks. The pharmacist will discuss with the participant the benefits of smoking cessation and will provide him or her with tailored behavioral and lifestyle strategies.
  To prevent nicotine withdrawal symptoms, the participant will be offered nicotine replacement therapy (NRT) The first follow-up session will be scheduled after 1 week of the participant's quit day and will take around 20 minutes. In this session, the pharmacist will determine the participant's smoking status and assess the NRT tolerability.
  • If the participant fails to quit smoking, the pharmacist will carefully review the participant's experience during the attempt to quit and will work through the identified problems
  Other Names: Participants will participate in a face-to-face 4-session program at the pharmacy delivered by the study pharmacist at 2-4-week intervals over 8 weeks.
  Arms: Intervention arm
Other: Control arm (i.e: regular care) — Participants in the control group will receive 5-10 minutes of unstructured brief smoking cessation advice by the pharmacist. In addition they will be provided with educational materials about smoking cessation and will be offered nicotine replacement therapy (NRT).
  Arms: Control arm

SUMMARY:
Thirty seven percent of adult male population smoke cigarettes in Qatar. The Global Youth Tobacco Survey also stated that 13.4% of male school students aged 13 to 15 years in Qatar smoke cigarettes. Smoking cessation is a key to reducing smoking related diseases and deaths. Health care providers are in an ideal position to encourage smoking cessation. Pharmacists are the most accessible health care providers and are uniquely situated to initiate behavior change among patients. Many western studies have shown that pharmacists can be successful in helping patients quit smoking. Studies demonstrating the effectiveness of pharmacist delivered smoking cessation programs are lacking in Qatar. This proposal aims to test the effect of a structured smoking cessation program delivered by trained ambulatory pharmacists in Qatar. A prospective, randomized, controlled trial will be conducted at 8 ambulatory pharmacies in Qatar. Participants will be randomly assigned to receive a 4-session face-to-face structured patient-specific smoking cessation program conducted by the pharmacist or 5 to 10 minutes of unstructured brief smoking cessation advice given by the pharmacist. Both groups will be offered nicotine therapy if feasible. The primary outcome of smoking cessation will be confirmed by exhaled carbon monoxide test at 12 months. If proven to be effective, this smoking cessation program will be considered as a model that Qatar and the region can apply to decrease smoking burden.

ELIGIBILITY:
Eligible participants are:

* patients aged 18 years and older who currently smoke one or more cigarettes daily for 7 days, are motivated to quit i.e.: in the preparation stage of the stage-of-change model, able to communicate in Arabic or English and are willing and capable of attending the scheduled sessions at the study pharmacies.

Exclusion criteria are:

* use of other nicotine or tobacco products
* current use or use in the last 30 days of quit smoking aids or medications
* plan to leave Qatar in the next 12 months
* presence of any major medical condition that would prevent use of the nicotine replacement therapy including hypersensitivity to the products, history of or recent myocardial infarction, life-threatening arrhythmias, severe or worsening angina, uncontrolled hypertension and temporomandibular joint disease (in case of nicotine gum)
* pregnancy
* psychiatric illness or other debilitating condition that would interfere with participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2013-02; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maguy S El Hajj, PharmD, Principal Investigator — Qatar University
Locations (2):
- Qatar (2):
  - Primary Health Corporation (PHC) pharmacies, Doha
  - Qatar Petroleum pharmacies, Doha

REFERENCES:
- [Derived] El Hajj MS, Kheir N, Al Mulla AM, Shami R, Fanous N, Mahfoud ZR. Effectiveness of a pharmacist-delivered smoking cessation program in the State of Qatar: a randomized controlled trial. BMC Public Health. 2017 Feb 20;17(1):215. doi: 10.1186/s12889-017-4103-4. PMID 28219367
- [Derived] El Hajj MS, Kheir N, Al Mulla AM, Al-Badriyeh D, Al Kaddour A, Mahfoud ZR, Salehi M, Fanous N. Assessing the effectiveness of a pharmacist-delivered smoking cessation program in the State of Qatar: study protocol for a randomized controlled trial. Trials. 2015 Feb 26;16:65. doi: 10.1186/s13063-015-0570-z. PMID 25885807

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between February 2013 and December 2014, the study pharmacists assessed 450 smokers for eligibility in the study. Of them, 361 (80.2%) met the study inclusion criteria. A total of 314 cigarette smokers consented to enroll in the study and were randomized into one of two study groups
Groups:
- Intervention Arm: Participants assigned to the intervention arm will participate in a face-to-face 4-session program at the pharmacy delivered by the study pharmacist at 2-4-week intervals over 8 weeks in addition to nicotine replacement therapy.
Period: 3 Month Outcome Measure
Arm/Group | Control Arm | Intervention Arm
Started | 147 | 167
Completed | 98 | 101
Not Completed | 49 | 66
Period: 6 Month Outcome Measure
Arm/Group | Control Arm | Intervention Arm
Started | 147 | 167
Completed | 99 | 100
Not Completed | 48 | 67
Period: 12 Month Outcome Measure
Arm/Group | Control Arm | Intervention Arm
Started | 147 | 167
Completed | 83 | 88
Not Completed | 64 | 79

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Arm | Intervention Arm | Total
Number analyzed (Participants) | 147 | 167 | 314
Age, Customized [Count of Participants; unit: Participants]
  18-29 years | 33 | 40 | 73
  30-39 years | 55 | 53 | 108
  40-49 years | 27 | 46 | 73
  50 years and above | 27 | 24 | 51
  Unknown | 5 | 4 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 143 | 164 | 307
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Nationality
  Participants
    Qatar | 36 | 25 | 61
    Egypt | 49 | 41 | 90
    Other countries | 60 | 96 | 156
    Unknown | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Self-reported 7-day Point Prevalence Abstinence
Description: Self-reported 7-day point prevalence abstinence, defined as having smoked no cigarettes for the previous 7 days
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 98 | 101
Participants | 26 | 31

2. Primary Outcome: Self-reported 30 Day Smoking Abstinence
Description: Self-reported 30-day point prevalence abstinence defined as having smoked no cigarettes in the last 30 days
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 98 | 101
Participants | 22 | 27

3. Primary Outcome: Self-reported Continuous Abstinence at 3 Months
Description: Self-reported continuous abstinence defined as having smoked no cigarettes since quit day
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 98 | 101
Participants | 21 | 25

4. Primary Outcome: Self-reported 7-day Point Prevalence Abstinence
Description: Defined as having smoked no cigarettes for the previous 7 days
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 99 | 100
Participants | 21 | 28

5. Primary Outcome: Self-reported 30-day Point Prevalence Abstinence
Description: Defined as having smoked no cigarettes in the last 30 days
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 99 | 100
Participants | 20 | 27

6. Primary Outcome: Self-reported Continuous Abstinence
Description: Defined as having smoked no cigarettes since quit day
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 99 | 100
Participants | 20 | 23

7. Primary Outcome: Self-reported 7-day Point Prevalence Abstinence
Description: Defined as having smoked no cigarettes for the previous 7 days
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 83 | 88
Participants | 14 | 21

8. Primary Outcome: Self-reported 30-day Point Prevalence Abstinence
Description: Defined as having smoked no cigarettes in the last 30 days
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 83 | 88
Participants | 14 | 21

9. Primary Outcome: Self-reported Continuous Abstinence
Description: Defined as having smoked no cigarettes since quit day at 12 months
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 83 | 88
participants | 14 | 21

10. Primary Outcome: Objective Smoking Abstinence
Description: Smoking abstinence as objectively verified by the CO exhaled test at 12 months
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 2 | 6
Participants | 2 | 6

11. Secondary Outcome: Health Related Quality of Life
Description: Mean change in health related quality of life score from baseline to 6 months for quitters vs. non quitters
Time Frame: 6 month
Population: Unfortunately patients didnt return at 6 months to fill the QOL questionnaire this is why we dont have data to report on this measure
Arm/Group | Control Arm | Intervention Arm
Number analyzed (Participants) | 0 | 0
Value | 0 | 0

ADVERSE EVENTS:
Arm/Group | Control Arm | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/147 | 0/167
Serious Adverse Events (participants affected / at risk) | 0/147 | 0/167
Other Adverse Events (participants affected / at risk) | 0/147 | 2/167
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Arm (N=147) | Intervention Arm (N=167)
Elevated Blood pressure (Cardiac disorders) | 0 (0) | 2 (2) — Elevated Blood pressure due to nicotine replacement therapy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No